CLINICAL TRIAL: NCT07127237
Title: Prucaloprida vs Bisacodyl as a Stimulant in Bowel Preparation for Video Colonoscopy in Adults: A Randomized Clinical Trial
Brief Title: Prucaloprida vs Bisacodyl as a Stimulant in Bowel Preparation for Video Colonoscopy in Adults
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital de Clínicas Dr. Manuel Quintela (Other)
Responsible Party: Principal Investigator, Ignacio Moratorio, Principal investigator, Hospital de Clínicas Dr. Manuel Quintela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HospitalCDMQ
Record Dates: First submitted 2025-06-23; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-06

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — Bisacodyl; prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bisacodyl (Experimental): On the day prior to the procedure, the group receiving bisacodyl will take 4 tablets (5 mg each) at 4:00 PM. Subsequently, at 6:00 PM, they will dissolve 3 sachets of PEG in 3 liters of water (1 sachet per liter) and ingest half of the preparation, that is, 1.5 liters over a period of 2 hours. At 10:00 PM, they will ingest the remaining 1.5 liters over another 2-hour period.
  Interventions: Drug: Bisacodyl 5 MG
- Prucaloprida (Experimental): On the day prior to the procedure, the group receiving prucalopride will take one 2 mg tablet at 4:00 PM. Subsequently, at 6:00 PM, they will dissolve 3 sachets of PEG in 3 liters of water (1 sachet per liter) and ingest half of the preparation-that is, 1.5 liters over a period of 2 hours. At 10:00 PM, they will ingest the remaining 1.5 liters over another 2-hour period.
  Interventions: Drug: Prucalopride 2mg

INTERVENTIONS:
Drug: Bisacodyl 5 MG — On the day prior to the procedure, the group receiving bisacodyl will take 4 tablets (5 mg each) at 4:00 PM. Subsequently, at 6:00 PM, they will dissolve 3 sachets of PEG in 3 liters of water (1 sachet per liter) and ingest half of the preparation, that is, 1.5 liters over a period of 2 hours. At 10:00 PM, they will ingest the remaining 1.5 liters over another 2-hour period.
  Arms: Bisacodyl
Drug: Prucalopride 2mg — On the day prior to the procedure, the group receiving prucaloprida will take 1 tablet (2 mg) at 4:00 PM. Subsequently, at 6:00 PM, they will dissolve 3 sachets of PEG in 3 liters of water (1 sachet per liter) and ingest half of the preparation, that is, 1.5 liters over a period of 2 hours. At 10:00 PM, they will ingest the remaining 1.5 liters over another 2-hour period.
  Arms: Prucaloprida

SUMMARY:
The objective of this randomized clinical trial is to compare prucalopride versus bisacodyl as a stimulant agent for bowel cleansing preparation prior to colonoscopy in patients undergoing the procedure at the Endoscopy Unit of the Hospital de Clínicas. The main research questions this study aims to answer are:

Is prucalopride superior or equivalent to bisacodyl as a stimulant agent for bowel cleansing preparation before colonoscopy? Is the tolerability of prucalopride better, equivalent, or worse compared to bisacodyl? The investigators will compare the standard bowel cleansing preparation using polyethylene glycol (PEG) in combination with either bisacodyl or prucalopride as the stimulant agent.

Participants will be randomized into two groups, both receiving the same base preparation with different stimulant agents.

DETAILED DESCRIPTION:
An analytical, experimental, prospective study will be conducted, specifically a triple-blind randomized clinical trial (blinding of the endoscopist, investigators, and statistician), comparing a bowel preparation regimen for colonoscopy using prucalopride versus bisacodyl.

Patients referred to the Digestive Endoscopy Unit of the Gastroenterology Department at the Hospital de Clínicas for colonoscopy (VCC) who meet the inclusion criteria will be invited to participate in the study. Referrals will include both hospitalized patients and outpatients from various clinic services.

Statistical Analysis Frequency tables and charts will be used to describe qualitative variables. Measures of central tendency and dispersion (mean ± standard deviation or median and interquartile range [IQR]) will be used for continuous variables depending on the distribution assessed by the Kolmogorov-Smirnov test.

Associations between qualitative variables will be analyzed using the Chi-square test or Fisher's exact test when expected frequencies are less than 5. If a statistically significant association is found, the strength of the association will be expressed using the Relative Risk (RR) and its corresponding 95% Confidence Interval (CI).

Differences between groups in normally distributed continuous variables will be analyzed using the Student's t-test for independent samples, and for non-normally distributed variables, the Mann-Whitney U test will be used.

Adenoma detection rate and cecal intubation rate will be calculated as the number of new cases (detection or cecal intubation) per total number of procedures performed. These rates will be expressed using the appropriate constant K based on the number of patients, along with their 95% CI. The comparison between groups will be performed using a test for comparison of independent proportions. A significance level of α = 0.05 will be established. Statistical analysis will be performed using STATA v.18.0.

Study Variables • Boston Bowel Preparation Scale (BBPS) Conceptual definition: A scale used to assess bowel cleanliness during colonoscopy.

Operational definition:

Score 0: unprepared colon segment with mucosa not visualized due to solid stool that cannot be cleared.

Score 1: portion of mucosa is seen, but other areas are obscured by staining, residual stool, and/or opaque liquid.

Score 2: minor residual staining or small fragments of stool, but mucosa is adequately visualized.

Score 3: entire mucosa is visible with no residual material. Type and scale: Qualitative, ordinal variable.

Categories:

Total score: 0-9. Adequate preparation: BBPS ≥ 2 in each colonic segment. Inadequate preparation: BBPS < 2 in any segment.

• Tolerance Conceptual definition: Refers to the presence or absence of specific symptoms during bowel preparation, including nausea, vomiting, abdominal pain or distension, headache, dizziness, fatigue, palpitations, and rectal bleeding.

Operational definition:

Good tolerance: ≤ 3 symptoms. Moderate tolerance: 4-5 symptoms. Poor tolerance: ≥ 6 symptoms. Type and scale: Qualitative, ordinal variable. Categories: Good, Moderate, Poor.

• Overall Adenoma Detection Rate (ADR) Conceptual definition: A quality indicator for colonoscopy. An ADR ≥ 25% is considered acceptable (≥ 30% in men and ≥ 20% in women).

Operational definition: Number of adenomas/adenocarcinomas (confirmed by histology) divided by the total number of colonoscopies performed, multiplied by 100.

Type and scale: Quantitative, continuous variable; ratio scale. Values: 0-100%.

• Overall Cecal Intubation Rate Conceptual definition: A quality indicator for colonoscopy. Considered acceptable if ≥ 95% in screening colonoscopies and ≥ 90% in other types of colonoscopies.

Operational definition: Number of colonoscopies where the ileocecal valve is visualized divided by the total number of colonoscopies performed, multiplied by 100.

Type and scale: Quantitative, continuous variable; ratio scale. Values: 0-100%.

Data Collection Method Patient Recruitment: All patients scheduled for colonoscopy at the Digestive Endoscopy Unit of the Hospital de Clínicas who meet the inclusion criteria will be invited to participate. Informed consent will be obtained after providing detailed explanations and resolving any questions.

Data Collection Tool: Individual standardized forms with closed-ended questions will be completed for each participant. One of the principal investigators will gather the necessary information to complete the baseline data collection form, including demographic data, medical history, and patient-reported experience with bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age.
* Without prior colonic surgical interventions.
* Who attend the Digestive Endoscopy service to undergo a colonoscopy.

Exclusion Criteria:

* Patients who voluntarily choose not to participate in the study.
* Pregnant women.
* Patients with rectocolonic resections and/or ileostomies.
* Inflammatory bowel disease.
* Inadequate bowel preparation in a previous colonoscopy.
* Suspected intestinal obstruction or perforation.
* Intestinal intussusception.
* Melena.
* Oral iron intake within the last 10 days.
* Emergency colonoscopies.
* Hypersensitivity to any component of the bowel preparation solutions.
* Chronic kidney disease on dialysis.
* Uncorrected severe electrolyte imbalances.
* Major psychiatric disorders.
* Low intellectual quotient.
* Severe constipation (≤ 1 bowel movement per week).
* Chronic diarrhea with high frequency (≥ 4 daily bowel movements of uniformly decreased consistency for more than 4 weeks).
* Decompensated cardiac diseases (ischemic heart disease, congestive heart failure, unstable angina, arrhythmias, and uncontrolled hypertension).
* Ascites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Boston scale | Periprocedural
  Scale used to evaluate the quality of bowel preparation during video colonoscopy. Score 0-9; adequate preparation (Boston ≥ 2 points in each colonic segment), inadequate preparation (Boston < 2 points in any of the segments).

SECONDARY OUTCOMES:
Tolerability of bowel preparation. Presence or absence of the following symptoms during bowel preparation: nausea, vomiting, abdominal pain or distension, headache, dizziness, fatigue, palpitations, and rectal bleeding. | Periprocedural
  Refers to the presence or absence of the following symptoms during bowel preparation: nausea, vomiting, abdominal pain or distension, headache, dizziness, fatigue, palpitations, and rectal bleeding. Tolerability will be assessed through a standardized questionnaire administered prior to colonoscopy.
Overall adenoma detection rate | Until the completion of the studies. Average 1 year
  Conceptual definition: A key quality indicator in colonoscopy. An overall adenoma detection rate ≥25% of procedures is considered acceptable (≥30% in men and ≥20% in women).
  Operational definition: Calculated as the number of adenomas/adenocarcinomas (confirmed by histological diagnosis) divided by the total number of colonoscopies performed, multiplied by 100.
Overall cecal intubation rate | Until the completion of the studies. Average 1 year.
  Conceptual definition: A quality indicator in colonoscopy. An acceptable rate is ≥95% for screening colonoscopies and ≥90% for other types of colonoscopies.
  Operational definition: Calculated as the number of colonoscopies in which the ileocecal valve is visualized, divided by the total number of colonoscopies performed, multiplied by 100.

IPD SHARING:
Plan to Share IPD: Yes
All collected data